CLINICAL TRIAL: NCT06012890
Title: Impact of Acquisition Automation on the Duration and Quality of Cardiac MRI Examinations
Brief Title: Performance of Acquisition Automation of Cardiac MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Carl Glessgen, Medical Doctor, Consultant, University Hospital, Geneva
Other Study IDs: 2023-01047
Record Dates: First submitted 2023-08-14; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Workflow; Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Automatic acquisition: Clinical MRI planning performed automatically by an AI-based software
  Interventions: Other: Automation of cardiac MRI acquisition
- Manual Acquisition: Clinical MRI planning performed manually by a specialized radiology technician

INTERVENTIONS:
Other: Automation of cardiac MRI acquisition — The intervention will consist of the automation of the cMRI examination.
  Groups: Automatic acquisition

SUMMARY:
For this study, cardiac MRI examinations performed will be prospectively included and realized either fully automatically or by a specialized radiology technician. The duration of the automated examinations will be compared to the duration of the manual examinations. The number of failed sequences in both study arms (automated and manual) will be recorded and the quality of the cardiac planes will be compared.

DETAILED DESCRIPTION:
The main hypothesis is that fully automated cardiac MRI protocols require shorter overall scan times than manually acquired, human-executed protocols. The objective will be to demonstrate that automating the examination allows to shorten the scan time, leading to increased patient comfort and clinical flexibility. The study's secondary objective will be to demonstrate the non-inferiority of the automated protocol compared to human acquisition in terms of resulting planning quality and error occurrence during slice planning.

Included patients will undergo clinical cMRI following international and national standards: only the acquisition strategy will vary. The investigators will successively recruit patients presenting for routine cardiac MRI. The acquisition strategy of the MRI - either automated or manual - will alternate to avoid comparison bias.

The MRI protocol will be the same for both arms and consists of standardized sequences acquired before and after contrast administration. Recruitment will be performed at a single location, in the radiology department. Patients will be recruited on a daily, consecutive basis during clinical practice.

No questionnaire will be used for this study. No biological material will be sampled. Observational data about the acquisition process, potential errors, and patient characteristics will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient presenting for morphologic and functional assessment of the myocardium by cardiac MRI.
* Research consent form obtained after information procedure.
* Complete cardiac MRI protocol performed.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Implantable cardiac device
* Incomplete cardiac examination due to early termination by the patient.
* Incomplete data on examination parameters (missing forms).
* Incompatible MRI protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population referred for morphological cardiac MRI, with consecutive patient sampling.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall scan time | Up to 12 months
  This study's primary endpoint will be the overall scan time, from first to last MRI image acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Glessgen, MD, Principal Investigator — Radiologist
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No